CLINICAL TRIAL: NCT04735874
Title: Vascular Health and Risk Factors in Children With Down Syndrome
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Boston Children's Hospital (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Adam Ware, MD, Assistant Professor, Pediatric Cardiology, University of Utah
Other Study IDs: 00127761
Record Dates: First submitted 2020-11-12; First posted 2021-02-03 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Down Syndrome; Cardiovascular Risk Factor; Atherosclerosis
Keywords: Down Syndrome; Cardiovascular Risk Factor; Atherosclerosis
MeSH Terms: conditions — Down Syndrome; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children ages 10.0 to 18.0
  Interventions: Other: Evaluate vascular disease risk factors in children with Down Syndrome; Other: Determine the associations between cardiovascular disease risk factors and markers of early atherosclerosis in children with Down Syndrome

INTERVENTIONS:
Other: Evaluate vascular disease risk factors in children with Down Syndrome — We will determine CV disease risk profiles in children with DS at our centers. We will compare these data to published national norms of children without DS. Risk factor data will include: anthropometric measures; blood pressure; history of congenital heart disease and associated surgery, sleep apnea, hypothyroidism, and cancer; fasting blood draw [lipid panel with subfractions (NMR), insulin, glucose, and CRP].
Other: Determine the associations between cardiovascular disease risk factors and markers of early atherosclerosis in children with Down Syndrome — We will perform PWV, CIMT, and CD studies in children with DS and compare these data to available data in children without DS. We will also perform multivariable analysis of the influence of combinations of CV disease risk factors on markers of early atherosclerosis in children with DS. Hypothesis: CV disease risk factors will correlate with markers of early atherosclerosis in children with DS but the associations between risk factors and markers of early atherosclerosis will differ between children with DS vs. the general population of children.

SUMMARY:
This is a prospective, multicenter, cross-sectional study to evaluate prevalence of vascular risk factors in children with Down Syndrome and to determine the association between vascular disease risk factors and objective markers of early atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* All children with Down Syndrome (10.0-18.0 years of age)
* Children with translocations and mosaicism
* Children with and without CHD

Exclusion Criteria:

* Patients with a history of hypoplastic arch, coarctation or catheter or surgical based aorta interventions
* Patients who are currently treated or have been treated with chemotherapy for cancer or a myeloproliferative disorder within 1 year of the study
* Participants whose parent/legally authorized representative (LAR) perceives the child is not able to cooperate with vascular imaging studies

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All children with DS (10.0-18.0 years of age) will be eligible, including those with translocations and mosaicism
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The difference in mean pulse wave velocity between children with Down syndrome and published national data in children without Down syndrome at one time point. | One day patient visit
  Pulse wave velocity (PWV) is a non-invasive imaging measure of arterial stiffness. Pulse wave velocity measures vascular stiffness by evaluating the time for a pressure wave to travel through the aorta. The velocity is determined by the elasticity and geometry of the vessel. PWV will be measured using a SphygmoCor device. With the participant in the supine position and ECG leads attached, the maximal pulsation of the right carotid and right femoral artery will be marked and measured from the suprasternal notch using a tape measure (carotid) and caliper (femoral). A tonometer will record the carotid and femoral impulses. The device calculates PWV as the difference in the carotid-to-distal path length divided by the difference in R-wave-to-waveform times (∆distance/∆time, m/sec). Measurements will be in triplicate and averaged. PWV can be completed in ~30 mins.

SECONDARY OUTCOMES:
The difference in mean carotid intimal medial thickness between children with Down syndrome and published national data in children without Down syndrome measured at 1 time point. | One day patient visit
  Carotid intimal medial thickness (CIMT) is a non-invasive imaging measure of carotid artery thickness. B-mode ultrasound with a high-resolution linear array vascular transducer will be used to record common, bulb, and internal CIMT.
Correlation of body mass index (BMI) anthropometric cardiovascular risk factors on PWV and CIMT in children with Down syndrome. | One day patient visit
  Height (centimeters) will be measured using standard stadiometers and weight (kilograms) using a calibrated scale available at each site. BMI (kg/m2) will be calculated and converted to age- and sex-matched Down Syndrome percentiles. Measured at 1 time point.
Correlation of waist circumference anthropometric cardiovascular risk factors on PWV and CIMT in children with Down syndrome. | One day patient visit
  Waist circumference will be measured at the top of the posterior iliac crest (NHANES standard) and normalized by calculating waist to height ratio. Measured at 1 time point.
Correlation of serologic cardiovascular risk factors include fasting lipid panel on PWV and CIMT in children with Down syndrome. | One day patient visit
  A fasting lipid profile will be obtained to measure total cholesterol, triglycerides, and HDL cholesterol. Trained pediatric phlebotomists will perform the blood draw after the participant has fasted ≥10 hours. A standard lipid profile will provide total cholesterol, HDL cholesterol, and triglycerides. LDL will be calculated using the Friedwald equation when triglycerides are <400 mg/dL. For triglycerides ≥400 mg/dl, LDL will be measured directly via a homogeneous enzymatic assay. Measured at 1 time point.
Correlation of serologic cardiovascular risk factors include lipoprotein on PWV and CIMT in children with Down syndrome. | One day patient visit
  Lipoprotein subfractions by NMR will be used to describe lipid particle number and size. These lipoprotein measurements likely estimate CV risk more accurately than a standard lipid profile alone. Lipoprotein sub-fractionation will be completed using proton NMR signals. Measured at 1 time point.
Correlation of serologic cardiovascular risk factors include insulin resistance on PWV and CIMT in children with Down syndrome. | One day patient visit
  Insulin resistance will be assessed by fasting serum glucose, hemoglobin A1C, and insulin level since diabetes (fasting glucose ≥126 mg/dL or hemoglobin A1C ≥6.5%) is a major risk factor. Measured at 1 time point.
Correlation of clinical cardiovascular risk factors on PWV and CIMT in children with Down syndrome. | One day patient visit
  A detailed personal history for congenital heart disease (CHD) and associated surgery, sleep apnea, hypothyroidism, and cancer will be obtained as all are common in the population with Down Syndrome and increase the risk for cardiovascular disease in adulthood. The fundamental CHD and associated surgery will be obtained from the medical records. The parent/LAR will be questioned and the medical record reviewed for a history of sleep apnea, hypothyroidism, and cancer (yes/no). Measured at 1 time point.

CONTACTS AND LOCATIONS:
Overall Officials: Adam L Ware, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ware AL, Miller DV, Porter CB, Edwards WD. Characterization of atrial morphology and sinus node morphology in heterotaxy syndrome: an autopsy-based study of 41 cases (1950-2008). Cardiovasc Pathol. 2012 Sep-Oct;21(5):421-7. doi: 10.1016/j.carpath.2011.12.007. Epub 2012 Jan 28. PMID 22285192
- [Background] Ware AL, Miller DV, Erickson LK, Menon SC. Marfan syndrome associated aortic disease in neonates and children: a clinical-morphologic review. Cardiovasc Pathol. 2016 Sep-Oct;25(5):418-22. doi: 10.1016/j.carpath.2016.06.002. Epub 2016 Jun 16. PMID 27479044
- [Background] Ware AL, Malmberg E, Delgado JC, Hammond ME, Miller DV, Stehlik J, Kfoury A, Revelo MP, Eckhauser A, Everitt MD. The use of circulating donor specific antibody to predict biopsy diagnosis of antibody-mediated rejection and to provide prognostic value after heart transplantation in children. J Heart Lung Transplant. 2016 Feb;35(2):179-85. doi: 10.1016/j.healun.2015.10.006. Epub 2015 Oct 8. PMID 26520246
- [Background] Ware AL, Tani LY, Weng HY, Wilkes J, Menon SC. Resource utilization and outcomes of infective endocarditis in children. J Pediatr. 2014 Oct;165(4):807-12.e1. doi: 10.1016/j.jpeds.2014.06.026. Epub 2014 Jul 23. PMID 25064162
- [Background] Ware AL, Young PC, Weng C, Presson AP, Minich LL, Menon SC. Prevalence of Coronary Artery Disease Risk Factors and Metabolic Syndrome in Children with Heart Disease. Pediatr Cardiol. 2018 Feb;39(2):261-267. doi: 10.1007/s00246-017-1750-2. Epub 2017 Oct 23. PMID 29058030
- [Background] Glasson EJ, Sullivan SG, Hussain R, Petterson BA, Montgomery PD, Bittles AH. The changing survival profile of people with Down's syndrome: implications for genetic counselling. Clin Genet. 2002 Nov;62(5):390-3. doi: 10.1034/j.1399-0004.2002.620506.x. PMID 12431254
- [Background] Head E, Phelan MJ, Doran E, Kim RC, Poon WW, Schmitt FA, Lott IT. Cerebrovascular pathology in Down syndrome and Alzheimer disease. Acta Neuropathol Commun. 2017 Dec 1;5(1):93. doi: 10.1186/s40478-017-0499-4. PMID 29195510
- [Background] Wilcock DM, Schmitt FA, Head E. Cerebrovascular contributions to aging and Alzheimer's disease in Down syndrome. Biochim Biophys Acta. 2016 May;1862(5):909-14. doi: 10.1016/j.bbadis.2015.11.007. Epub 2015 Nov 26. PMID 26593849
- [Background] Sobey CG, Judkins CP, Sundararajan V, Phan TG, Drummond GR, Srikanth VK. Risk of Major Cardiovascular Events in People with Down Syndrome. PLoS One. 2015 Sep 30;10(9):e0137093. doi: 10.1371/journal.pone.0137093. eCollection 2015. PMID 26421620
- [Background] Yla-Herttuala S, Luoma J, Nikkari T, Kivimaki T. Down's syndrome and atherosclerosis. Atherosclerosis. 1989 Apr;76(2-3):269-72. doi: 10.1016/0021-9150(89)90110-x. PMID 2525042
- [Background] Brattstrom L, Englund E, Brun A. Does Down syndrome support homocysteine theory of arteriosclerosis? Lancet. 1987 Feb 14;1(8529):391-2. doi: 10.1016/s0140-6736(87)91772-7. No abstract available. PMID 2880201
- [Background] Murdoch JC, Rodger JC, Rao SS, Fletcher CD, Dunnigan MG. Down's syndrome: an atheroma-free model? Br Med J. 1977 Jul 23;2(6081):226-8. doi: 10.1136/bmj.2.6081.226. PMID 141966
- [Background] Alexander M, Petri H, Ding Y, Wandel C, Khwaja O, Foskett N. Morbidity and medication in a large population of individuals with Down syndrome compared to the general population. Dev Med Child Neurol. 2016 Mar;58(3):246-54. doi: 10.1111/dmcn.12868. Epub 2015 Aug 18. PMID 26282180
- [Background] Expert Panel on Integrated Guidelines for Cardiovascular Health and Risk Reduction in Children and Adolescents; National Heart, Lung, and Blood Institute. Expert panel on integrated guidelines for cardiovascular health and risk reduction in children and adolescents: summary report. Pediatrics. 2011 Dec;128 Suppl 5(Suppl 5):S213-56. doi: 10.1542/peds.2009-2107C. Epub 2011 Nov 14. No abstract available. PMID 22084329
- [Background] Vis JC, Winter MM, Weijerman ME, et al. Down syndrome Congenital heart defects in Down syndrome Prevalence of congenital heart defects. 2019;53(5):1-22
- [Background] Parra P, Costa R, de Asua DR, Moldenhauer F, Suarez C. Atherosclerotic Surrogate Markers in Adults With Down Syndrome: A Case-Control Study. J Clin Hypertens (Greenwich). 2017 Feb;19(2):205-211. doi: 10.1111/jch.12890. Epub 2016 Aug 6. PMID 27495829
- [Background] Vis JC, Duffels MG, Winter MM, Weijerman ME, Cobben JM, Huisman SA, Mulder BJ. Down syndrome: a cardiovascular perspective. J Intellect Disabil Res. 2009 May;53(5):419-25. doi: 10.1111/j.1365-2788.2009.01158.x. Epub 2009 Feb 18. PMID 19228275
- [Background] Zhu JL, Hasle H, Correa A, Schendel D, Friedman JM, Olsen J, Rasmussen SA. Survival among people with Down syndrome: a nationwide population-based study in Denmark. Genet Med. 2013 Jan;15(1):64-9. doi: 10.1038/gim.2012.93. Epub 2012 Aug 9. PMID 22878506
- [Background] Foerste T, Sabin M, Reid S, Reddihough D. Understanding the causes of obesity in children with trisomy 21: hyperphagia vs physical inactivity. J Intellect Disabil Res. 2016 Sep;60(9):856-64. doi: 10.1111/jir.12259. Epub 2016 Mar 3. PMID 26936540
- [Background] van Gameren-Oosterom HB, van Dommelen P, Schonbeck Y, Oudesluys-Murphy AM, van Wouwe JP, Buitendijk SE. Prevalence of overweight in Dutch children with Down syndrome. Pediatrics. 2012 Dec;130(6):e1520-6. doi: 10.1542/peds.2012-0886. Epub 2012 Nov 12. PMID 23147968
- [Background] Adelekan T, Magge S, Shults J, Stallings V, Stettler N. Lipid profiles of children with Down syndrome compared with their siblings. Pediatrics. 2012 Jun;129(6):e1382-7. doi: 10.1542/peds.2011-1262. Epub 2012 May 14. PMID 22585768
- [Background] Rouch L, Cestac P, Sallerin B, Andrieu S, Bailly H, Beunardeau M, Cohen A, Dubail D, Hernandorena I, Seux ML, Vidal JS, Hanon O. Pulse Wave Velocity Is Associated With Greater Risk of Dementia in Mild Cognitive Impairment Patients. Hypertension. 2018 Nov;72(5):1109-1116. doi: 10.1161/HYPERTENSIONAHA.118.11443. PMID 30354804
- [Background] Mattace-Raso FU, van der Cammen TJ, Hofman A, van Popele NM, Bos ML, Schalekamp MA, Asmar R, Reneman RS, Hoeks AP, Breteler MM, Witteman JC. Arterial stiffness and risk of coronary heart disease and stroke: the Rotterdam Study. Circulation. 2006 Feb 7;113(5):657-63. doi: 10.1161/CIRCULATIONAHA.105.555235. PMID 16461838
- [Background] Rodrigues AN, Coelho LC, Goncalves WL, Gouvea SA, Vasconcellos MJ, Cunha RS, Abreu GR. Stiffness of the large arteries in individuals with and without Down syndrome. Vasc Health Risk Manag. 2011;7:375-81. doi: 10.2147/VHRM.S21273. Epub 2011 Jun 9. PMID 21731889
- [Background] Kulsum-Mecci N, Goss C, Kozel BA, Garbutt JM, Schechtman KB, Dharnidharka VR. Effects of Obesity and Hypertension on Pulse Wave Velocity in Children. J Clin Hypertens (Greenwich). 2017 Mar;19(3):221-226. doi: 10.1111/jch.12892. Epub 2016 Aug 11. PMID 27511880
- [Background] Khan SS, Ning H, Wilkins JT, Allen N, Carnethon M, Berry JD, Sweis RN, Lloyd-Jones DM. Association of Body Mass Index With Lifetime Risk of Cardiovascular Disease and Compression of Morbidity. JAMA Cardiol. 2018 Apr 1;3(4):280-287. doi: 10.1001/jamacardio.2018.0022. PMID 29490333
- [Background] Kotlyarevska K, Wolfgram P, Lee JM. Is waist circumference a better predictor of insulin resistance than body mass index in U.S. adolescents? J Adolesc Health. 2011 Sep;49(3):330-3. doi: 10.1016/j.jadohealth.2010.12.008. Epub 2011 May 4. PMID 21856529
- [Background] Hatch-Stein JA, Zemel BS, Prasad D, Kalkwarf HJ, Pipan M, Magge SN, Kelly A. Body Composition and BMI Growth Charts in Children With Down Syndrome. Pediatrics. 2016 Oct;138(4):e20160541. doi: 10.1542/peds.2016-0541. Epub 2016 Sep 14. PMID 27630073
- [Background] Bertapelli F, Pitetti K, Agiovlasitis S, Guerra-Junior G. Overweight and obesity in children and adolescents with Down syndrome-prevalence, determinants, consequences, and interventions: A literature review. Res Dev Disabil. 2016 Oct;57:181-92. doi: 10.1016/j.ridd.2016.06.018. Epub 2016 Jul 19. PMID 27448331
- [Background] Freedman DS, Khan LK, Serdula MK, Dietz WH, Srinivasan SR, Berenson GS. The relation of childhood BMI to adult adiposity: the Bogalusa Heart Study. Pediatrics. 2005 Jan;115(1):22-7. doi: 10.1542/peds.2004-0220. PMID 15629977
- [Background] de Koning L, Merchant AT, Pogue J, Anand SS. Waist circumference and waist-to-hip ratio as predictors of cardiovascular events: meta-regression analysis of prospective studies. Eur Heart J. 2007 Apr;28(7):850-6. doi: 10.1093/eurheartj/ehm026. Epub 2007 Apr 2. PMID 17403720
- [Background] Sharma AK, Metzger DL, Daymont C, Hadjiyannakis S, Rodd CJ. LMS tables for waist-circumference and waist-height ratio Z-scores in children aged 5-19 y in NHANES III: association with cardio-metabolic risks. Pediatr Res. 2015 Dec;78(6):723-9. doi: 10.1038/pr.2015.160. Epub 2015 Sep 2. PMID 26331767
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- [Background] Poirier P, Giles TD, Bray GA, Hong Y, Stern JS, Pi-Sunyer FX, Eckel RH; American Heart Association; Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Obesity and cardiovascular disease: pathophysiology, evaluation, and effect of weight loss: an update of the 1997 American Heart Association Scientific Statement on Obesity and Heart Disease from the Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Circulation. 2006 Feb 14;113(6):898-918. doi: 10.1161/CIRCULATIONAHA.106.171016. Epub 2005 Dec 27. PMID 16380542
- [Background] Flynn JT, Kaelber DC, Baker-Smith CM, Blowey D, Carroll AE, Daniels SR, de Ferranti SD, Dionne JM, Falkner B, Flinn SK, Gidding SS, Goodwin C, Leu MG, Powers ME, Rea C, Samuels J, Simasek M, Thaker VV, Urbina EM; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BLOOD PRESSURE IN CHILDREN. Clinical Practice Guideline for Screening and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2017 Sep;140(3):e20171904. doi: 10.1542/peds.2017-1904. Epub 2017 Aug 21. PMID 28827377
- [Background] Yang Q, Rasmussen SA, Friedman JM. Mortality associated with Down's syndrome in the USA from 1983 to 1997: a population-based study. Lancet. 2002 Mar 23;359(9311):1019-25. doi: 10.1016/s0140-6736(02)08092-3. PMID 11937181
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Akhuemonkhan E, Lazo M. Association between family history of diabetes and cardiovascular disease and lifestyle risk factors in the United States population: The 2009-2012 National Health and Nutrition Examination Survey. Prev Med. 2017 Mar;96:129-134. doi: 10.1016/j.ypmed.2016.12.015. Epub 2016 Dec 19. PMID 28007493
- [Background] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of abnormal lipid levels among youths --- United States, 1999-2006. MMWR Morb Mortal Wkly Rep. 2010 Jan 22;59(2):29-33. PMID 20094024
- [Background] Duncan GE. Prevalence of diabetes and impaired fasting glucose levels among US adolescents: National Health and Nutrition Examination Survey, 1999-2002. Arch Pediatr Adolesc Med. 2006 May;160(5):523-8. doi: 10.1001/archpedi.160.5.523. PMID 16651496
- [Background] Saaddine JB, Fagot-Campagna A, Rolka D, Narayan KM, Geiss L, Eberhardt M, Flegal KM. Distribution of HbA(1c) levels for children and young adults in the U.S.: Third National Health and Nutrition Examination Survey. Diabetes Care. 2002 Aug;25(8):1326-30. doi: 10.2337/diacare.25.8.1326. PMID 12145229
- [Background] Ford ES, Li C, Zhao G, Mokdad AH. Concentrations of low-density lipoprotein cholesterol and total cholesterol among children and adolescents in the United States. Circulation. 2009 Mar 3;119(8):1108-15. doi: 10.1161/CIRCULATIONAHA.108.816769. Epub 2009 Feb 16. PMID 19221218
- [Background] Loprinzi P, Cardinal B, Crespo C, Brodowicz G, Andersen R, Sullivan E, Smit E. Objectively measured physical activity and C-reactive protein: National Health and Nutrition Examination Survey 2003-2004. Scand J Med Sci Sports. 2013 Mar;23(2):164-70. doi: 10.1111/j.1600-0838.2011.01356.x. Epub 2011 Aug 3. PMID 21812825
- [Background] Urbina EM, Williams RV, Alpert BS, Collins RT, Daniels SR, Hayman L, Jacobson M, Mahoney L, Mietus-Snyder M, Rocchini A, Steinberger J, McCrindle B; American Heart Association Atherosclerosis, Hypertension, and Obesity in Youth Committee of the Council on Cardiovascular Disease in the Young. Noninvasive assessment of subclinical atherosclerosis in children and adolescents: recommendations for standard assessment for clinical research: a scientific statement from the American Heart Association. Hypertension. 2009 Nov;54(5):919-50. doi: 10.1161/HYPERTENSIONAHA.109.192639. Epub 2009 Sep 3. PMID 19729599
- [Background] Iwakiri T, Yano Y, Sato Y, Hatakeyama K, Marutsuka K, Fujimoto S, Kitamura K, Kario K, Asada Y. Usefulness of carotid intima-media thickness measurement as an indicator of generalized atherosclerosis: findings from autopsy analysis. Atherosclerosis. 2012 Dec;225(2):359-62. doi: 10.1016/j.atherosclerosis.2012.10.033. Epub 2012 Oct 12. PMID 23092826
- [Background] Park MH, Skow A, De Matteis S, Kessel AS, Saxena S, Viner RM, Kinra S. Adiposity and carotid-intima media thickness in children and adolescents: a systematic review. BMC Pediatr. 2015 Oct 16;15:161. doi: 10.1186/s12887-015-0478-5. PMID 26475608
- [Background] Urbina EM. Abnormalities of vascular structure and function in pediatric hypertension. Pediatr Nephrol. 2016 Jul;31(7):1061-70. doi: 10.1007/s00467-015-3188-1. Epub 2015 Aug 15. PMID 26275663
- [Background] Doyon A, Kracht D, Bayazit AK, Deveci M, Duzova A, Krmar RT, Litwin M, Niemirska A, Oguz B, Schmidt BM, Sozeri B, Querfeld U, Melk A, Schaefer F, Wuhl E; 4C Study Consortium. Carotid artery intima-media thickness and distensibility in children and adolescents: reference values and role of body dimensions. Hypertension. 2013 Sep;62(3):550-6. doi: 10.1161/HYPERTENSIONAHA.113.01297. Epub 2013 Jul 1. PMID 23817494
- [Background] Croymans DM, Sanchez A, Barth JD, Roberts CK. Carotid intima-media thickness, dietary intake, and cardiovascular phenotypes in adolescents: relation to metabolic syndrome. Metabolism. 2010 Apr;59(4):533-9. doi: 10.1016/j.metabol.2009.08.016. Epub 2009 Oct 20. PMID 19846177
- [Background] Mittelman SD, Gilsanz P, Mo AO, Wood J, Dorey F, Gilsanz V. Adiposity predicts carotid intima-media thickness in healthy children and adolescents. J Pediatr. 2010 Apr;156(4):592-7.e2. doi: 10.1016/j.jpeds.2009.10.014. Epub 2009 Dec 14. PMID 20004913
- [Background] White D, Place R, Michael T, Hoffman E, Gordon PM, Visich P. The Relationship between Coronary Artery Disease Risk Factors and Carotid Intima-Media Thickness in Children. J Pediatr. 2017 Nov;190:38-42. doi: 10.1016/j.jpeds.2017.07.034. Epub 2017 Sep 11. PMID 28912051
- [Background] Vergeer M, Zhou R, Bots ML, Duivenvoorden R, Koglin J, Akdim F, Mitchel YB, Huijgen R, Sapre A, de Groot E, Sijbrands EJ, Pasternak RC, Gagne C, Marais AD, Ballantyne CM, Isaacsohn JL, Stalenhoef AF, Kastelein JJ. Carotid atherosclerosis progression in familial hypercholesterolemia patients: a pooled analysis of the ASAP, ENHANCE, RADIANCE 1, and CAPTIVATE studies. Circ Cardiovasc Imaging. 2010 Jul;3(4):398-404. doi: 10.1161/CIRCIMAGING.109.909655. Epub 2010 May 21. PMID 20494942
- [Background] Giannini C, Diesse L, D'Adamo E, Chiavaroli V, de Giorgis T, Di Iorio C, Chiarelli F, Mohn A. Influence of the Mediterranean diet on carotid intima-media thickness in hypercholesterolaemic children: a 12-month intervention study. Nutr Metab Cardiovasc Dis. 2014 Jan;24(1):75-82. doi: 10.1016/j.numecd.2013.04.005. Epub 2013 Jun 25. PMID 23809150
- [Background] Mikola H, Pahkala K, Niinikoski H, Ronnemaa T, Viikari JSA, Jula A, Juonala M, Raitakari OT. Cardiometabolic Determinants of Carotid and Aortic Distensibility From Childhood to Early Adulthood. Hypertension. 2017 Aug;70(2):452-460. doi: 10.1161/HYPERTENSIONAHA.117.09027. Epub 2017 Jun 26. PMID 28652463
- [Background] Leone N, Ducimetiere P, Gariepy J, Courbon D, Tzourio C, Dartigues JF, Ritchie K, Alperovitch A, Amouyel P, Safar ME, Zureik M. Distension of the carotid artery and risk of coronary events: the three-city study. Arterioscler Thromb Vasc Biol. 2008 Jul;28(7):1392-7. doi: 10.1161/ATVBAHA.108.164582. Epub 2008 Apr 17. PMID 18421001
- [Background] Yang EY, Chambless L, Sharrett AR, Virani SS, Liu X, Tang Z, Boerwinkle E, Ballantyne CM, Nambi V. Carotid arterial wall characteristics are associated with incident ischemic stroke but not coronary heart disease in the Atherosclerosis Risk in Communities (ARIC) study. Stroke. 2012 Jan;43(1):103-8. doi: 10.1161/STROKEAHA.111.626200. Epub 2011 Oct 27. PMID 22033999
- [Background] Khoury M, Manlhiot C, Dobbin S, Gibson D, Chahal N, Wong H, Davies J, Stearne K, Fisher A, McCrindle BW. Role of waist measures in characterizing the lipid and blood pressure assessment of adolescents classified by body mass index. Arch Pediatr Adolesc Med. 2012 Aug;166(8):719-24. doi: 10.1001/archpediatrics.2012.126. PMID 22473884
- [Background] Jeyarajah EJ, Cromwell WC, Otvos JD. Lipoprotein particle analysis by nuclear magnetic resonance spectroscopy. Clin Lab Med. 2006 Dec;26(4):847-70. doi: 10.1016/j.cll.2006.07.006. PMID 17110242
- [Background] Greenland S, Robins JM. Estimation of a common effect parameter from sparse follow-up data. Biometrics. 1985 Mar;41(1):55-68. PMID 4005387
- [Background] Schwarzer G. meta: An R Package for Meta-Analysis. R News. 2007;7:40-45
- See also: R Core Team (2018). R: A language and environment for statistical computing. R Foundation for Statistical Computing. Published 2018. — https://www.r-project.org/